CLINICAL TRIAL: NCT05373199
Title: A Trial Comparing the Pharmacodynamics and Pharmacokinetics of BC Combo THDB0207 and Lantus® and Humalog® in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Collaborators: Tonghua Dongbao Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CT047-ADO05
Record Dates: First submitted 2022-05-04; First posted 2022-05-13 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucose Clamp Technique; Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Intervention Model Description: Three-period crossover
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BC Combo THDB0207 (Experimental): Single administration of BC Combo THDB0207
  Interventions: Drug: Euglycemic clamp with BC Combo THDB0207
- Lantus® (Active Comparator): Single administration of Lantus®
  Interventions: Drug: Euglycemic clamp with Lantus®
- Humalog® (Active Comparator): Single administration of Humalog®
  Interventions: Drug: Euglycemic clamp with Humalog®

INTERVENTIONS:
Drug: Euglycemic clamp with BC Combo THDB0207 — Administration of a single dose of BC Combo THDB0207 during an euglycemic clamp procedure.
  Arms: BC Combo THDB0207
Drug: Euglycemic clamp with Lantus® — Administration of a single dose of Lantus® during an euglycemic clamp procedure.
  Arms: Lantus®
Drug: Euglycemic clamp with Humalog® — Administration of a single dose of Humalog® during an euglycemic clamp procedure.
  Arms: Humalog®

SUMMARY:
This is a randomised, double-blind, three-period crossover euglycaemic clamp trial comparing pharmacokinetics and pharmacodynamics of BC Combo THDB0207 and Lantus® and Humalog® in subjects with type 1 diabetes.

Each subject will be randomly allocated to one of the 6 treatment sequences and will be administered single subcutaneous doses of BC Combo THDB0207, Lantus®, and Humalog® at three separate dosing visits.

Subjects will come in a fasted state to the clinical trial centre in the morning of each dosing day and stay at the clinical trial centre until the 24-hour clamp procedures have been terminated. Patients will return to the clinical trial centre for outpatient blood sampling visits for analysis of BC449 excipient until 144 hours after each dosing.

DETAILED DESCRIPTION:
Subjects will attend the study site in the morning in a fasted state and will be connected to an automated glucose clamp device (ClampArt). Prior to dose administration plasma glucose will be stabilised at a target level of 100 mg/dL by means of an intravenous infusion of glucose or insulin. IMP administration will be done by an unblinded person by means of subcutaneous injections in the abdominal wall.

Following each dosing a euglycaemic glucose clamp procedure will be carried out for up to 24 hours.

The pharmacodynamic assessment will be based on the time course of glucose infusion rate (GIR) and plasma glucose.

Plasma insulin concentrations will be measured using a specific validated bioanalytical method differentiating concentrations of insulin glargine, of its main metabolites insulin glargine-M1 and insulin glargine-M2, and of insulin lispro. Pharmacokinetic assessments will be based on total insulin (INS) concentration (insulin glargine + insulin glargine-M1 + insulin glargine-M2 + insulin lispro).

The investigation of PK properties of the BC449 excipient after dosing with BC Combo THDB0207 will be based on blood samples collected during the clamp procedure and at daily outpatient visits until 144 hours after dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) for ≥ 12 months
* HbA1c ≤8.5%
* Total insulin dose of < 1.2 U/kg/day
* BMI between 20.0 and 29.9 kg/m2 (both inclusive)
* Treated with insulin regimen for ≥ 12 months prior to screening
* Using multiple dosing insulin therapy (MDI) with basal and bolus insulin or insulin pump therapy (continuous subcutaneous insulin infusion, CSII)
* Fasting C-peptide <= 0.30 nmol/L

Exclusion Criteria:

* Known or suspected hypersensitivity to the IMPs or any of the excipients or to any component of the IMP formulation.
* Type 2 diabetes mellitus
* Use of oral antidiabetic drugs (OADs) and/or GLP-1 receptor agonists (e.g. exenatide, liraglutide)
* Receipt of any medicinal product in clinical development within 30 days or at least 5 half-lives of the related substances and their metabolites (whichever is longer) before randomisation in this trial
* Clinically significant abnormal screening laboratory tests, as judged by the Investigator considering the underlying disease
* Clinically relevant comorbidity, capable of constituting a risk for the subject when participating in the trial or of interfering with the interpretation of data
* Systolic blood pressure < 90 mmHg or >139 mmHg and/or diastolic blood pressure < 50 mmHg or > 89 mmHg (one repeat test will be acceptable in case of suspected white-coat hypertension)
* Heart rate at rest outside the range of 50-90 beats per minute.
* More than one episode of severe hypoglycaemia with seizure, coma or requiring assistance of another person during the past 6 months or hypoglycaemia unawareness as judged by the investigator
* Women of childbearing potential who are not using a highly effective contraceptive method.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
AUCGIR 0-6h | From t=0 to t=6 hours after IMP administration
  Area under the glucose infusion rate curve until 6 hours after dosing of BC Combo THDB0207 and Lantus®
AUCGIR 6-24h | From t=6 to t=24 hours after IMP administration
  Area under the glucose infusion rate curve from 6 hours to 24 hours after dosing of BC Combo THDB0207 and Humalog®

SECONDARY OUTCOMES:
AUCGIR 0-last | From t=0 to t=24 hours after IMP administration
  Area under the glucose infusion rate curve from 0 hours until the end of clamp
AUCGIR 0-4h | From t=0 to t=4 hours after IMP administration
  Area under the glucose infusion rate curve from 0 hours until 4 hours
GIRmax | From t=0 to t=24 hours
  Maximum glucose infusion rate
tGIRmax | From t=0 to t=24 hours
  Time to maximum glucose infusion rate
tonset of action | From t=0 to t=24 hours after IMP administration
  Time until Plasma Glucose (PG) has decreased by at least 5 mg/dL from the baseline PG value.
AUCINS 0-6h | From t=0 to t=6 hours after IMP administration
  Area under the insulin concentration-time curve from 0 hours until 6 hours
AUCINS 0-24h | From t=0 to t=24 hours after IMP administration
  Area under the insulin concentration-time curve from 0 hours until 24 hours
AUCINS 6-24h | From t=6 to t=24 hours after IMP administration
  Area under the insulin concentration-time curve from 6 hours until 24 hours
AUCINS 4-12h | From t=4 to t=12 hours after IMP administration
  Area under the insulin concentration-time curve from 4 hours until 12 hours
AUCINS 0-4h | From t=0 to t=4 hours after IMP administration
  Area under the insulin concentration-time curve from 0 hours until 4 hours
AUCINSlast | From t=0 to t=24 hours
  Area under the insulin concentration-time curve from t=0 to the last measured insulin concentration above LLOQ
Cmax INS | From t=0 to t=24 hours after IMP administration
  Maximum insulin concentration
RBA | From t=0 to t=24 hours after IMP administration
  Relative bioavailability of BC Combo THDB0207 vs Humalog®
AUCBC 0-12h | From t=0 to t=12 hours after IMP administration
  Area under the BC449 concentration-time curve from 0 hours until 12 hours
AUCBC 0-24h | From t=0 to t=24 hours after IMP administration
  Area under the BC449 concentration-time curve from 0 hours until 24 hours
AUCBC 0-last | From t=0 to t=144 hours after IMP administration
  Area under the BC449 concentration-time curve from t=0 to the last measured BC449 concentration above LLOQ
Adverse Events | From the first IMP administration to the follow-up visit (i.e. up to 11 weeks)
  Incidence of Adverse Events
Local tolerability | From the first IMP administration to the follow-up visit (i.e. up to 11 weeks)
  Incidence of injection site reactions

CONTACTS AND LOCATIONS:
Overall Officials: Marc Stoffel, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany